CLINICAL TRIAL: NCT01468532
Title: Phase I/II Trial to Establish the Safety and Preliminary Efficacy of the Combination of Docetaxel, Prednisone, and SOM 230 (Pasireotide) in Metastatic Castrate Resistant Prostate Cancer (CRPC).
Brief Title: Docetaxel, Prednisone, and Pasireotide in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-031; NCI-2011-03216 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-10-25; First posted 2011-11-09 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; pasireotide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, receptor agonist) (Experimental): Patients receive pasireotide IM, 40 mg on day 1, docetaxel 75mg/m2 IV over 1 hour, and prednisone 5mg PO BID continuously. Courses with docetaxel repeat every 21 days and courses with pasireotide repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: pasireotide; Drug: prednisone

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: pasireotide — Given IM
  Other Names: SOM230
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra

SUMMARY:
This phase I/II trial studies the side effects and best dose of pasireotide and to see how well it works when given together with docetaxel and prednisone in treating patients with metastatic hormone-resistant prostate cancer. Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pasireotide may inhibit the secretion of hormones. Giving pasireotide together with docetaxel and prednisone may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) level of SOM 230 (pasireotide) in combination with docetaxel and prednisone.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination in metastatic castration-resistant prostate cancer (CRPC).

II. To evaluate preliminary efficacy of the combination of SOM 230 and docetaxel and prednisone as defined by response rates (measurable and prostate-specific antigen [PSA]), time to progression (TTP) and overall survival (OS).

III. To evaluate the pharmacokinetics (PK) of the combination. IV. To assess the pharmacodynamic (PD) effects of the combination as seen by baseline levels of and changes in insulin-like growth factor (IGF)-1, serum chromogranin A (SCA), and neuron specific enolase (NSE), and to associate them with TTP and OS.

V. To assess the pretherapy circulating tumor cell (CTC) counts and change in CTC after therapy, and to associate them with TTP and OS.

OUTLINE: This is a phase I dose-escalation study of pasireotide followed by a phase II study.

Patients receive pasireotide intramuscularly (IM) on day 1, docetaxel intravenously (IV) over 1 hour, and prednisone orally (PO) twice daily (BID) continuously. Courses with docetaxel repeat every 21 days and courses with pasireotide repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma with metastasis, and objective progression or rising PSA despite androgen deprivation therapy and antiandrogen withdrawal when applicable; patients with rising PSA must demonstrate a rising trend with 2 successive elevations at a minimum interval of 1 week; a minimum PSA of 5 ng/ml or new areas of bony metastases on bone scan are required for patients with no measurable disease; no minimum PSA requirement for patients with measurable disease
* Patient must not have received any prior chemotherapy for metastatic disease; all patients must be documented to be castrate with a testosterone level < 0.5 ng/ml; luteinizing hormone-releasing hormone (LHRH) agonist therapy must be continued, if required to maintain castrate levels of testosterone; patients must be off antiandrogens for a minimum of 4 weeks for flutamide and 6 weeks for bicalutamide or nilutamide
* Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy 12 weeks or more
* Absolute neutrophil (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hgb) > 9 g/dL
* Serum bilirubin =< 2 x upper limit of normal (ULN)
* Serum transaminases activity =< 3 x ULN, with the exception of serum transaminases (< 5 x ULN) if the patient has liver metastases
* Serum creatinine =< 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN; NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Patients must be advised of the importance of using effective birth control measures during the course of the study
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information

Exclusion Criteria:

* Prior treatment with any cytotoxic chemotherapy, radiation, immunotherapy, or any investigational drug within the preceding 4 weeks
* Patients who have undergone major surgery within 4 weeks prior to study enrollment
* Chronic treatment with immunosuppressive agents except steroids
* Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years
* Patients with uncontrolled diabetes mellitus, which is defined as a hemoglobin A1C > 8% on therapy or > 7% without therapy, or a fasting plasma glucose > 1.5 ULN; Note: at the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted
* Patients with symptomatic cholelithiasis
* Patients who have congestive heart failure (New York Heart Association [NYHA] Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment
* QT-related exclusion criteria:
* Patients with baseline QTc > or = 470 msec
* History of syncope or family history of idiopathic sudden death
* Sustained or clinically significant cardiac arrhythmias
* Patients with risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
* Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes or Parkinson's disease), human immunodeficiency virus (HIV), cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Concomitant medication(s) known to prolong the QT interval
* Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (enzyme-linked immunosorbent assay [ELISA] and Western blot)
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* Severely impaired lung function
* Any active (acute or chronic) or uncontrolled infection/ disorders
* Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide long-acting release (LAR) formulations
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Men and any female partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation and for additional 2 months after finishing therapy; should a patient's sexual partner become pregnant or suspect she is pregnant while patient is participating in this study, he should inform the treating physician immediately

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulka Vaishampayan, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy, Receptor Agonist): Patients receive pasireotide IM on day 1, docetaxel IV over 1 hour, and prednisone PO BID continuously. Courses with docetaxel repeat every 21 days and courses with pasireotide repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  docetaxel: Given IV
  pasireotide: Given IM
  prednisone: Given PO
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 65 [49 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Pasireotide in Combination With Docetaxel and Prednisone by the Occurrence of Adverse Events and the Associated Grade Per NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: To identify the maximum tolerated dose (MTD) of pasireotide, The occurrence rate of binary endpoints (eg, specific types of toxicity at a certain dose level and severity grade, response, etc) will be described by point estimates and exact 90% confidence intervals (CIs) for proportions using Wilson's method.
Time Frame: Up to day 57
Measure: Number; unit: mg
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
mg | 60

2. Secondary Outcome: The Number of Patients With Toxicity as Assessed Via NCI CTCAE Version 4.0
Description: The count of patients who experience a given type and grade of toxicity as assessed via NCI CTCAE version 4.0
Time Frame: On days 1, 8, 15, 22, 29, 36 43, 50 and 57
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
Participants
  Abdominal pain grade 1 | 1
  Agitation grade 1 | 1
  Alkaline phosphatase increased grade 3 | 3
  Allergic reaction grade 1 | 1
  Alopecia grade 1 | 1
  Alopecia grade 2 | 1
  Anemia grade 1 | 4
  Anemia grade 3 | 4
  Anorexia grade 1 | 6
  Anorexia grade 2 | 1
  Arthritis grade 1 | 2
  Aspartate aminotransferase increased grade 2 | 1
  Aspartate aminotransferase increased grade 3 | 1
  Back pain grade 1 | 3
  Back pain grade 2 | 1
  Bladder infection grade 2 | 1
  Blood and lymphatic system disorders-Other grade 1 | 1
  Bruising grade 1 | 1
  Cardiac disorders - Other, specify grade 1 | 1
  Cataract grade 1 | 1
  Chills grade 1 | 4
  Cholesterol high grade 1 | 5
  Conjunctivitis grade 2 | 1
  Constipation grade 1 | 4
  Cough grade 1 | 2
  Cough grade 2 | 1
  Creatinine increased grade 1 | 1
  Dehydration grade 2 | 2
  Dehydration grade 3 | 1
  Depression grade 1 | 2
  Diarrhea grade 1 | 10
  Diarrhea grade 2 | 2
  Diarrhea grade 3 | 1
  Dizziness grade 1 | 8
  Dry mouth grade 1 | 2
  Dry skin grade 1 | 2
  Dysgeusia grade 1 | 1
  Dysgeusia grade 2 | 4
  Dyspnea grade 1 | 6
  Ear and labyrinth disorders-Other, specify grade 1 | 1
  Edema limbs grade 1 | 1
  Edema limbs grade 2 | 1
  EKG QT corrected interval prolong grade 1 | 1
  EKG QT corrected interval prolong grade 2 | 1
  EKG QT corrected interval prolong grade 3 | 1
  Eye disorders - Other, specify grade 1 | 2
  Fatigue grade 1 | 6
  Fatigue grade 2 | 7
  Fatigue grade 3 | 1
  Fever grade 1 | 1
  Flank pain grade 1 | 1
  Flu like symptoms grade 1 | 2
  Flushing grade 1 | 2
  Gastroesophageal reflux disease grade 1 | 3
  Gastroesophageal reflux disease grade 2 | 1
  Gastrointestinal disorders -Other, specify grade 1 | 7
  Generalized muscle weakness grade 1 | 5
  Generalized muscle weakness grade 2 | 2
  Headache grade 1 | 1
  Hearing impaired grade 1 | 1
  Heart failure grade 1 | 1
  Hematuria grade 1 | 2
  Hematuria grade 2 | 1
  Hoarseness grade 1 | 1
  Hot flashes grade 1 | 3
  Hyperglycemia grade 1 | 3
  Hyperglycemia grade 2 | 1
  Hyperglycemia grade 3 | 10
  Hyperkalemia grade 2 | 1
  Hypertension grade 2 | 5
  Hypertension grade 3 | 5
  Hypertriglyceridemia grade 1 | 3
  Hypertriglyceridemia grade 3 | 1
  Hypoalbuminemia grade 3 | 1
  Hypocalcemia grade 1 | 1
  Hypocalcemia grade 3 | 1
  Hypokalemia grade 2 | 2
  Hypomagnesemia grade 1 | 1
  Hypomagnesemia grade 2 | 1
  Hyponatremia grade 3 | 4
  Hypophosphatemia grade 3 | 3
  Hypotension grade 3 | 1
  Hypothyroidism grade 1 | 1
  Infusion related reaction grade 2 | 1
  Infusion site extravasation grade 2 | 1
  Injection site reaction grade 1 | 1
  Insomnia grade 1 | 1
  Localized edema grade 1 | 1
  Lymphedema grade 1 | 1
  Lymphocyte count decreased grade 1 | 1
  Lymphocyte count decreased grade 3 | 7
  Lymphocyte count decreased grade 4 | 1
  Mucositis oral grade 2 | 1
  Muscle weakness lower limb grade 1 | 2
  Musculoskeletal and connective tissue dis. grade 1 | 5
  Myalgia grade 1 | 1
  Nail discoloration grade 1 | 2
  Nail discoloration grade 2 | 1
  Nail loss grade 1 | 1
  Nail ridging grade 1 | 2
  Nasal congestion grade 1 | 1
  Nausea grade 1 | 10
  Nausea grade 2 | 1
  Nervous system disorders - Other grade 1 | 1
  Neutrophil count decreased grade 3 | 10
  Neutrophil count decreased grade 4 | 6
  Otitis externa grade 2 | 1
  Pain grade 1 | 2
  Pain in extremity grade 2 | 1
  Pelvic pain grade 1 | 1
  Penile infection grade 1 | 1
  Penile pain grade 1 | 1
  Peripheral sensory neuropathy grade 1 | 7
  Peripheral sensory neuropathy grade 2 | 4
  Platelet count decreased grade 1 | 1
  Rash acneiform grade 1 | 6
  Rash acneiform grade 2 | 1
  Rectal pain grade 1 | 2
  Renal and urinary disorders - Other grade 1 | 1
  Renal and urinary disorders - Other grade 2 | 2
  Respiratory, thoracic and mediastinal dis. grade 3 | 1
  Serum amylase increased grade 4 | 1
  Sinus disorder grade 1 | 1
  Sinusitis grade 2 | 1
  Skin and subcutaneous tissue disorders grade 1 | 9
  Skin and subcutaneous tissue disorders grade 2 | 1
  Skin infection grade 4 | 1
  Sore throat grade 1 | 3
  Thromboembolic event grade 3 | 1
  Toothache grade 1 | 1
  Tremor grade 1 | 1
  Upper respiratory infection grade 1 | 2
  Upper respiratory infection grade 2 | 1
  Upper respiratory infection grade 3 | 1
  Urinary frequency grade 1 | 4
  Urinary tract infection grade 2 | 4
  Urinary tract infection grade 3 | 1
  Urinary tract obstruction grade 2 | 1
  Vomiting grade 1 | 4
  Watering eyes grade 1 | 1
  Weight loss grade 1 | 1
  Weight loss grade 2 | 6
  Weight loss grade 3 | 1
  Wheezing grade 1 | 1
  White blood cell decreased grade 3 | 11
  White blood cell decreased grade 4 | 3

3. Secondary Outcome: Measurements of Tumor Using Response Evaluation Criteria In Solid Tumors (RECIST) Criteria Before and After Treatment With the Combination of Pasireotide in Combination With Docetaxel
Description: Percentage of participants responding to treatment by measurements of tumor using Response Evaluation Criteria In Solid Tumors (RECISTv1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR, before and after treatment with the combination of pasireotide in combination with docetaxel
Time Frame: Every 12 weeks for the first 36 weeks and then every 16 weeks thereafter up to 100 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
percentage of participants | 44.4 [27.2 to 63.1]

4. Secondary Outcome: Percentage Prostate-specific Antigen (PSA) Change Noted
Description: Percentage change of prostate-specific antigen (PSA) decline or increase noted
Time Frame: On days 1, 22, 43
Measure: Median (Full Range); unit: percentage change of PSA from day 1
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
percentage change of PSA from day 1
  from day 1 to day 22 | -18.52 [-70.97 to 147.40]
  from day 1 to day 43 | -31.49 [-88.14 to 88.89]

5. Secondary Outcome: Time to Progression (TTP)
Description: Time from Treatment start date to Progression (TTP) Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Every 3 months for the first 9 months on study then every 4 months after the first 9 months on study, up to 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
months | 7.2 [3.8 to 8.2]

6. Secondary Outcome: Overall Survival (OS)
Description: Time from Treatment start date to date of death or last follow-up.
Time Frame: Every 3 months for the first 9 months on study then every 4 months after the first 9 months on study
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
months | 18.3 [15.0 to 29.7]

7. Secondary Outcome: Pharmacokinetics (PK) of SOM230
Description: Pharmacokinetics (PK) of SOM230 measured in the bloodstream (in ng/ml) at days 29, 57, and 85.
Time Frame: Predosing/end of infusion/2, 3, 4 ,7, 24 and 48 hours after start of docetaxel; Day 43; predosing for docetaxel and pasireotide/end of infusion/2, 3, 4, 7, 24 hours day 44/48 hours day 45 after start of infusion; days 29, 57, and 85 prior to pasireotide
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
ng/ml
  Level at day 29 | 15.4 [4.75 to 46.1]
  Level at day 57 | 14.9 [5.15 to 34.2]
  Level at day 85 | 14.5 [3.38 to 35.2]

8. Secondary Outcome: Measurement of Levels of IGF-1, Serum Chromogranin A (SCA), and Neuron Specific Enolase (NSE), the Change Between Time Points Pre-therapy, Post-therapy
Description: Measurement of levels of IGF-1, serum chromogranin A (SCA), and neuron specific enolase (NSE), the change between time points (day 22 and day 43) from day 1 as measured in percent change.
Time Frame: Baseline and days 22 and 43
Measure: Median (Full Range); unit: percent change of biomarker from day 1
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
percent change of biomarker from day 1
  IGF-1 day 1 to day 22 | -47.74 [-81.67 to 420.00]
  IGF-1 day 1 to day 43 | -65.64 [-76.85 to 9200.00]
  SCA day 1 to day 22 | -25.36 [-82.17 to 76.09]
  SCA day 1 to day 43 | -21.43 [-92.21 to 173.91]
  NSE day 1 to day 22 | -17.00 [-82.32 to 294.44]
  NSE day 1 to day 43 | 8.00 [-70.12 to 61.11]

9. Secondary Outcome: Measurements of CTC Counts, the Change Between Time-points Pre-therapy, Post-therapy
Description: Measurements of CTC counts, the change between time-points (day 22 and day 43) from day 1 as measured in percent change.
Time Frame: Baseline and days 22 and 43
Measure: Median (Full Range); unit: percent change of CTC from day 1
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
Number analyzed (Participants) | 18
percent change of CTC from day 1
  CTC from day 1 to day 22 | -5.50 [-1424.00 to 93.00]
  CTC from day 1 to day 43 | -29.50 [-1446.00 to 19.00]

ADVERSE EVENTS:
Time Frame: Any All-Cause Mortality, Serious, or Other (Not Including Serious) adverse event occurring after the patient has provided informed consent and until 4 weeks after the patient has stopped study participation must be reported, an average of 2 years.
Description: These will be followed per IND requirements (if applicable) as well as per sponsor requirements and WSU IRB requirements.
Arm/Group | Treatment (Chemotherapy, Receptor Agonist)
All-Cause Mortality (participants affected / at risk) | 13/18
Serious Adverse Events (participants affected / at risk) | 14/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Receptor Agonist) (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (Blood and lymphatic system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Receptor Agonist) (N=18)
Fatigue (General disorders) | 17 (35)
Diarrhea (Gastrointestinal disorders) | 13 (17)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT01468532/Prot_SAP_000.pdf